Virtual Reality Pain Neuroscience Education for middle school students

USD- IRB-20-129,

NCT04470375

# The University of South Dakota Child's Assent

## What is a research study?

A research study is something like a science project at school, but harder to do. When doctors and scientists want to learn more about a treatment, they have to test it on people to see if the treatment helps people and to make sure it does not hurt them.

## Why do you want me to be in this study?

The people who are running this study think finding out how children like yourself learn about pain in a virtual reality environment might help other children. That is why we are asking you to help us test the virtual reality pain education. You do not have to be in the study if you do not want to be

#### What do I have to do?

If you choose to be in this study, researchers Dr. Kory Zimney or Adriaan Louw

- Will have you fill out some questions about yourself and your current knowledge and beliefs about pain.
- They will then set you up with virtual reality googles and have you watch about a 30-minute virtual reality session teaching you about pain.
- When you are done with the virtual reality session they will ask you the same questions about your knowledge and beliefs about pain.
- You will be with the researchers about 1 hour to complete both sets of questions before and after along with viewing the virtual reality session.
- Sometimes people feel dizzy or get an upset stomach watching virtual reality, you can stop if you get any of these symptoms or anything else that does not feel right to you.

You can ask any question you want before you decide if you want to be in this research study. The researchers will answer your questions.

## What if I do not want to be in this study?

You do not have to be in this study even if your parents say it is OK. If you do not want to be in the study, the researcher will not force you to be in it. If you decide to be in the study, but change your mind, you can stop being in the study.

If you do not want to be in the study, or if you change your mind, just tell the researcher.

## Could I be hurt if I am in the study?

A small number of people (about 1 in 4,000) do not do well while viewing virtual reality. They may get dizzy, blackout, eye or muscle twitching, or other strange symptoms.

If you feel sick or are afraid that something is wrong with you, tell an adult at once.

\*\*\*\*\*\*\*\*\*

| Now I think I know about the study and what it means. Here is what I decided: | |
|---|---|
| <ul><li>□ NO, I do not want to be in the study.</li><li>□ OK, I will be in the study.</li></ul> | |
| Your name (printing is OK) Date | |
| I certify that this study and the procedures involved have been explained to in terms he/sh could understand and that he/she freely assented to participate in this study. | ıe |
| Signature of Person Obtaining Assent Date/time | |
| Name (print) | |